CLINICAL TRIAL: NCT00050713
Title: Sirolimus Therapy in Idiopathic and Lupus Membranous Nephropathy
Brief Title: Sirolimus Therapy for Idiopathic and Lupus Membranous Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030071; 03-DK-0071
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-07-07

CONDITIONS: Membranous Glomerulonephritis; Lupus Membranous Nepropathy
Keywords: Kidney Disease; Glomerulonephritis; Lupus Nephritis; Nephrotic Syndrome; Hyperlipidemia
MeSH Terms: conditions — Glomerulonephritis, Membranous; Kidney Diseases; Glomerulonephritis; Lupus Nephritis; Nephrotic Syndrome; Hyperlipidemias | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
This study will evaluate the safety and effectiveness of a new immunosuppressive drug, sirolimus, in reducing the amount of protein in the urine in patients with membranous nephropathy. This condition involves damage to the walls of tiny blood vessel filters in the kidneys called glomeruli, which allows blood proteins to leak into the urine. Patients have low blood protein levels and high blood cholesterol. Some patients may have leg swelling, impaired kidney function, blood vessel and heart disease, and a risk of emboli (blood clots that travel to the lungs). Drugs currently used to treat membranous nephropathy vary in their effectiveness among patients and can cause severe side effects.

The Food and Drug Administration has approved sirolimus for suppressing the immune system of patients who have had a kidney transplant to reduce the risk of organ rejection. The drug does not have certain side effects that have caused problems for patients treated with other immunosuppressants, such as: prednisone (weight gain, round face, diabetes, weak and fractured bones, and cataracts); cyclophosphamide (fertility problems, bladder injury and bladder cancer, and other cancers); chlorambucil (fertility problems, seizures, acute leukemia, and other cancers); and cyclosporine (kidney toxicity, increased facial hair, and seizures).

Patients 13 years of age or older with idiopathic membranous nephropathy or lupus membranous nephropathy may be eligible for this study. Candidates must have completed at least one month of treatment with a stable dose of angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs). They will be screened with a medical history, physical examination, blood tests, skin test for exposure to tuberculosis, and an examination for infection, cancers, and other conditions that can cause membranous nephropathy.

Participants will take sirolimus once a day for 1 year, except for the first day of treatment, when they will take three doses to quickly bring their blood levels of the drug up to a therapeutic level. They will undergo evaluations at the NIH in Bethesda, Maryland, at baseline (before starting treatment) and again at 1- to 4-month intervals during the study. In addition, they will have blood tests every week for the first month and every 2 weeks for the second month; then blood and urine tests once a month for the next 10 months of treatment and then every 4 months for a 12-month period after treatment stops. These tests will evaluate drug side effects and the response to therapy, and will determine if the therapeutic benefits persist long-term when treatment stops.

Patients will also be asked to have optional kidney function tests during the baseline evaluation and at the end of the follow-up period to measure kidney filtration and blood flow rates. Those who participate will be given fluids and other substances by vein to accurately measure kidney function. They will then have blood and urine samples collected about four times over a 1-hour period after drinking fluids to increase urine output.

Patients who experience a substantial increase in proteinuria or substantial decrease in kidney function during the course of treatment will stop taking sirolimus and be taken off the study.

DETAILED DESCRIPTION:
This is a phase 2 trial to evaluate the safety and effectiveness of a new immunosuppressive drug, sirolimus, in patients with idiopathic and lupus membranous nephropathy. Patients (age greater than or equal to 13 years) will be invited to participate if they have persistent nephrotic range proteinuria despite standard treatment with an angiotensin converting enzyme inhibitor or an angiotensin receptor blocker for at least one month, unless intolerant. These individuals are at risk for renal function deterioration as well as cardiovascular and thrombo-embolic complications of the nephrotic syndrome. Renal function, the degree of proteinuria and side effects will be monitored closely throughout the study. Physiologic measures of glomerular function will be examined at study entry and at the conclusion of the trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Ability and willingness to provide informed consent (adults greater than or equal to 18 years) or assent (children greater than or equal to 13 years) to all aspects of the study after full information is provided.

Nephrotic range proteinuria that persists for at least 3 months.

Nephrotic range proteinuria that persists despite angiotensin antagonist therapy (ACE inhibitor or ARB) for at least on month, unless intolerant. If patients have not started ACE inhibitor therapy before they are referred to NIH, we plan to start lisinopril 5 mg daily. We will advance the dose of ACE inhibitor as tolerated. Nephrotic range proteinuria, defined as 24 hour urine protein excretion greater than or equal to 3.5 g/d, must be documented in at least two 24 hour urine collections obtained during the month prior to initiating sirolimus. Incomplete urine collections (based on inadequate creatinine excretion) will be excluded.

Renal biopsy must reveal typical changes of membranous nephropathy by light and electron microscopy.

SLE as defined by the presence of at least 4 criteria established by the American Rheumatism Association (Lupus Membranous Nephropathy) or no evidence of a secondary form of membranous nephropathy (Idiopathic Membranous Nephropathy).

EXCLUSION CRITERIA:

Intolerance to sirolimus or prior use of sirolimus for membranous nephropathy.

Estimated GFR less than 30 mL/min/1.73(2) (determined by the 5 variable version of the MDRD Study prediction equation).

Immunosuppressive medications or experimental medications of any type during the two-month period prior to initiating sirolimus, with the following two exceptions:

First, patients with lupus membranous nephropathy are permitted to have received modest doses of corticosteroids (no more than the equivalent of prednisone 10mg/day) for control of extra-renal manifestations of SLE during the two-month period prior to starting sirolimus treatment.

Second, patients with worsening nephrotic syndrome (urine protein excretion rate doubles +/or serum albumin decreases by greater than or equal to 1.0 g/ dL to less than 2.5 g/dL on at least 2 determinations during or following a previous immunosuppressive treatment) should fulfill the following criteria:

a) should be off prednisone for at least 2 weeks before performing the baseline evaluation and starting sirolimus (if the patient has idiopathic membranous nephropathy): b) should be on low-dose corticosteroids (no more than the equivalent of prednisone 10 mg/day) for at least 2 weeks before performing the baseline evaluation and starting sirolimus (if the patient lupus membranous nephropathy); c) should be off cyclosporine for at least 2 weeks before performing the baseline evaluation and starting sirolimus; d) should be off cyclophosphamide, chlorambucil, azathioprine and mycophenolate mofetil for at least 4 weeks before performing the baseline evaluation and starting sirolimus;

Children less than 13.0 years.

Active acute or chronic infection requiring antimicrobial therapy or serious viral infection (e.g. HIV, hepatitis, herpes zoster). Patients with a reactive PPD must have completed a 6 to 12 month course of isoniazid as recommended by an infectious disease consultant. Patients with a non-reactive PPD and non-reactive anergy panel must complete a 6 to 12 month course of isoniazid if recommended by an infectious disease consultant.

Pregnant women, nursing mothers or individuals (men and women) not practicing birth control.

Uncontrolled hypertension, defined as BP greater than 140/90 on greater than 25% of measurements. Blood pressures will be measured 3 times at each clinic visit after the patient has sat quietly for at least 5 minutes. Thus at least 6 BP determinations will be recorded prior to initiating sirolimus therapy.

Chronic liver disease sufficiently severe to impair sirolimus metabolism; this would include prolonged pro-thrombin time. Patients with abnormal liver function tests will be evaluated by the Hepatology Consult Service to determine whether protocol participation is appropriate.

Basal thrombocytopenia less than 100,000 cells/microliters or absolute neutrophil count less than 2000 cells/microliters or hematocrit less than 30.

Cancer diagnosis or cancer recurrence within the preceding 5 years, excluding basal cell carcinoma of the skin.

Routine use of NSAIDS, defined as NSAID use more than two doses a week.

Clinically significant medical conditions, which in the opinion of the investigators, could increase the subject s risk of participating in the study or could confound the interpretation of the results of the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2002-12-17; Primary Completion 2007-08-27 (Actual); Study Completion 2007-08-27 (Actual)

PRIMARY OUTCOMES:
The number of patients who are in 1) complete remission or 2) complete or partial remission. | 12 months after starting sirolimus

SECONDARY OUTCOMES:
The number of patients who are in Complete or Partial Remission or Limited Response. | 12 months after starting sirolimus
Frequency of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Austin, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Farquhar MG, Saito A, Kerjaschki D, Orlando RA. The Heymann nephritis antigenic complex: megalin (gp330) and RAP. J Am Soc Nephrol. 1995 Jul;6(1):35-47. doi: 10.1681/ASN.V6135. PMID 7579068
- [Background] Kerjaschki D, Neale TJ. Molecular mechanisms of glomerular injury in rat experimental membranous nephropathy (Heymann nephritis). J Am Soc Nephrol. 1996 Dec;7(12):2518-26. doi: 10.1681/ASN.V7122518. PMID 8989729
- [Background] McMillan JI, Riordan JW, Couser WG, Pollock AS, Lovett DH. Characterization of a glomerular epithelial cell metalloproteinase as matrix metalloproteinase-9 with enhanced expression in a model of membranous nephropathy. J Clin Invest. 1996 Feb 15;97(4):1094-101. doi: 10.1172/JCI118502. PMID 8613533